CLINICAL TRIAL: NCT05989451
Title: Adaptation of Individual Dialectical Behavior Therapy Intervention for Transdiagnostic Treatment of Emotional Disorders in Two Medical Centers: a Randomized Controlled Trial
Brief Title: Adaptation of Individual Dialectical Behavior Therapy Intervention for Transdiagnostic Treatment of Emotional Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Senior Visiting Staff, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 112-2314-B-195 -007 -MY3
Record Dates: First submitted 2023-07-13; First posted 2023-08-14 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Anxiety Disorder; Depressive Disorder
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as Usual (TAU) (No Intervention): Treatment-as-usual (TAU) is a naturalistic treatment condition as delivered in current daily practice by psychiatrists in the medical services in Taiwan. TAU typically includes prescription and monitoring of antidepressant and/or anxiolytic medication, psychological treatment (this may include empathic listening and/or supportive counselling, psychoeducation, etc), or a combination of both. Patients in the TAU condition already receiving any of the aforementioned treatments are informed they will continue to receive as usual the services received before enrollment in the study.
- Transdiagnostic Adapted DBT plus TAU (Experimental): The modified DBT protocol, developed by the principal investigator and co-investigators, which will be offered in an individual therapy format. It consists of 12 weekly individual sessions, each lasting 50-60 minutes. It is made based on the manual (Linehan 2015), retaining the essence of DBT (Linehan 1993), and remain dialectically focused. Each session focuses on specific skills within that content of modules.
  Interventions: Behavioral: Dialectical behavior therapy (DBT)

INTERVENTIONS:
Behavioral: Dialectical behavior therapy (DBT) — The modified DBT protocol, developed by the principal investigator and co-investigators, will be offered in an individual therapy format. It consists of 12 weekly individual sessions, each lasting 50-60 minutes. It is made based on the manual, retaining the essence of DBT and remaining dialectically focused. Each session focuses on specific skills within the context of modules.
  Arms: Transdiagnostic Adapted DBT plus TAU

SUMMARY:
Anxiety and depressive disorders, referred to as emotional disorders, have high rates of prevalence, recurrence, and functional impairment. Transdiagnostic psychotherapy targeting shared features of these disorders has recently emerged. Dialectical behavior therapy (DBT) for the transdiagnostic treatment of emotional disorders is a promising approach, as results of preliminary studies for use in a broad range of mental disorders are encouraging. Since there is a lack of research on transdiagnostic psychotherapy in Taiwan, the investigators thus propose this 3-year randomized controlled trial to test the efficacy of a modified DBT for the treatment of transdiagnostic emotional disorders and to further evaluate whether the efficacy of modified DBT differs in the specific emotional disorders. The investigators expect that patients with emotional disorders receiving modified DBT are more likely to improve clinical outcomes, functioning, and quality of life.

DETAILED DESCRIPTION:
Anxiety and depressive disorders, referred to as emotional disorders, have high rates of prevalence, recurrence, and functional impairment. Transdiagnostic psychotherapy targeting shared features of these disorders has recently emerged. Dialectical behavior therapy (DBT) for the transdiagnostic treatment of emotional disorders is a promising approach, as results of preliminary studies for use in a broad range of mental disorders are encouraging. Since there is a lack of research on transdiagnostic psychotherapy in Taiwan, the investigators thus propose this 3-year randomized controlled trial to test the efficacy of a modified DBT for the treatment of transdiagnostic emotional disorders and to further evaluate whether the efficacy of modified DBT differs in the specific emotional disorders. This 3-year intervention trial has a randomized, controlled, two-center, and single-blinded design with two parallel groups. The trial will be conducted in the psychiatry departments of two medical centers, employing identical protocols. Participants will be recruited and randomly allocated 1:1 to one of two study arms. The modified DBT protocol in an individual therapy format consists of 12 weekly individual sessions, each lasting 50 minutes. A minimum of 250 participants will be included based on sample size estimation. Assessments will take place before the start of the trial, at the end of the trial, and at a 3-month follow-up. Primary outcomes will be the severity of depression and anxiety, rated by blind assessors. Secondary outcomes include disorder-specific symptoms, disorder severity, functional impairment, quality of life, and emotion regulation biases. The investigators will also examine the treatment mechanisms and treatment processes.

ELIGIBILITY:
Inclusion Criteria:

1. Mandarin Chinese-language proficiency sufficient to complete study questionnaire
2. A current diagnosis of depressive or anxiety disorder as diagnosed from a SCAN interview

Exclusion Criteria:

1. Intellectual disability
2. Substance use disorder in the past three months
3. Bipolar disorder
4. Psychotic disorder
5. Organic brain disorder
6. Acute suicidality or a history of frequent or recent suicide attempts
7. Recent (past six weeks) change in psychiatric medication or unwillingness to maintain a stable dosage of medication during study participation
8. Had received five or more sessions of CBT in the past five years or unwilling to stop concurrent psychotherapy for an emotional disorder
9. Any mental or physical condition requiring hospital admission
10. Another medical condition likely to prevent participation in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change of total score of Hamilton Depression Scale-17 item (HAMD-17) | at baseline, at 20 weeks, at 32 week
  Hamilton Depression Scale-17 item is an interview-based instrument for rating the overall levels of severity of the symptoms of depression and the response to treatment. Each item is rated from 0 to 4 or 0 to 2; the scores correspond to increases in severity. Total scores range from 0 to 52.
Change of total score of Hamilton Anxiety Scale (HAM-A) | at baseline, at 20 weeks, at 32 week
  HAM-A comprises 14 items with each item being divided into five grades, based on a scale of 0 to 4, with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change of total score of Clinical Global Impressions-Severity (CGI-S) and Improvement (CGI-I) | at baseline, at 20 weeks, at 32 week
  CGI-S (severity): the current condition of the patient on a scale of 1-7 (1 being normal, and 7 being among the most severely ill patients). CGI-I (improvement): the degree of improvement, as perceived by the clinician, since the start of treatment of a scale of 1-7, 1 being very much improved, and 7 being very much worse.

SECONDARY OUTCOMES:
Change of total score of Depression, Anxiety, and Stress Scales (DASS-21) | at baseline, at 20 weeks, at 32 week
  DASS-21 is a self-report measure of depression, anxiety and stress. Each seven-item scale has four response options ranging from 0 (do not apply to me at all) to 3 (apply to me much, or most of the time). Higher scores on each scale indicate higher depression, anxiety, and distress.
Change of total score of Patient Health Questionnaire-9 items (PHQ-9) | at baseline, at 20 weeks, at 32 week
  PHQ-9 is a nine-item self-rated questionnaire to measure the severity of depressive symptoms corresponding to the DSM-V criteria of MDD. Each item of the PHQ-9 requires a response on a 4-point scale, ranging from 0 (never) to 3 (nearly everyday), for a total score ranging from 0 to 27, with higher scores indicating increased likelihood for major depressive disorder.
Change of total score of Generalized Anxiety Disorder-7 items (GAD-7) | at baseline, at 20 weeks, at 32 week
  GAD-7 is a seven-item self-rated questionnaire to assess the severity of generalized anxiety disorder according to DSM-IV diagnostic criteria. Each item is scored on a four-point Likert scale (0-3) with total scores ranging from 0 to 21 with higher scores reflecting greater anxiety severity.
Change of total score of Panic Disorder Severity Scale- Self Rating (PDSS-SR) | at baseline, at 20 weeks, at 32 week
  PDSS-SR is a self-reported instrument to rate the overall severity of panic disorder. It consists of 7 items coded on a 5-point ordinal scale (0-4), in which higher scores indicate a more severe panic attack.
Change of total score of Penn State Worry Questionnaire (PSWQ) | at baseline, at 20 weeks, at 32 week
  PSWQ has been widely used as a self-report measure of worry and GAD in most treatment outcome studies of GAD. It has 16 items and each item is rated on a scale from 1 ('not at all typical of me') to 5 ('very typical of me'). Total score indicate greater levels of pathological worry.
Change of total score of Short Form Social Interaction Anxiety (SIAS) | at baseline, at 20 weeks, at 32 week
  The Social Interaction Anxiety Scale (SIAS) is companion measures developed for social anxiety. It is among the most commonly used tool for assessing social anxiety and the outcome of psychosocial therapy. Short-form SIAS is the self-report scale with items rated on a 5-point Likert-type scale with values ranging from 0 "Not at all characteristic or true of me" to 4 "Extremely characteristic or true of me". Higher scores indicate more severe social anxiety.
Change of total score of Short Form Social Phobia Scale (SPS) | at baseline, at 20 weeks, at 32 week
  The Social Phobia Scale (SPS) is companion measures developed for social anxiety. It is among the most commonly used tool for assessing social anxiety and the outcome of psychosocial therapy. Short-form SPS is the self-report scale with items rated on a 5-point Likert-type scale with values ranging from 0 "Not at all characteristic or true of me" to 4 "Extremely characteristic or true of me". Higher scores indicate more severe social anxiety.
Change of total score of Difficulties in Emotional Regulation Scale (DERS) | at baseline, at 20 weeks, at 32 week
  DERS including 36 items which assess difficulties regulating emotion across six domains, will be used to assess emotional dysregulation. Items are rated on a scale of 1 ("almost never ") to 5 ("almost always"). Higher scores indicate more difficulty in emotion regulation.
Change of total score of International Positive and Negative Affect Schedule-Short Form (PANAS-SF) | at baseline, at 20 weeks, at 32 week
  The 10-item I-PANAS-SF includes five items measuring positive affect (PA) and five items measuring negative affect (NA). Responses were provided on a 5-point Likert scale ranging from 1 (never) to 5 (always). The higher scores on both PA and NA items indicate the tendency to experience a positive and negative mood.
Change of total score of Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q SF) | at baseline, at 20 weeks, at 32 week
  It evaluates overall enjoyment and satisfaction with physical health, mood, work, household and leisure activities, social and family relationships, daily functioning, sexual life, economic status, overall well-being and medications. Items are rated on a 5-point scale ('not at all or never' to 'frequently or all the time'), which higher scores indicate better enjoyment and satisfaction with life.
Change of total score of The Work and Social Adjustment Scale (WSAS) | at baseline, at 20 weeks, at 32 week
  WSAS was developed to measure the functional impairment resulting from a health problem. Each item is rated on a 9-point Likert scale from 0 (no impairment) to 8 (very severe impaired). Total scores range from 0 to 40; scores of <10 indicate a subclinical condition, 10 to 20 significant functional impairment but less severe clinical symptomatology, and ≥20 moderately severe psychopathology.
Change of total score of skills subscale (DSS) of the DBT Ways of Coping Checklist (DBT-WCCL) | at baseline, at 20 weeks, at 32 week
  DBT Skills Subscale (DSS; 38 items), which assesses adaptive coping responses. Participants rate how often they have used each strategy in the past month using a 4-point Likert-type scale from 0 (never used) to 3 (regularly used).Higher scores indicate more frequent use of these skills.

OTHER OUTCOMES:
Change of diagnosis of Schedules for Clinical Assessment in Neuropsychiatry (SCAN) | at baseline, at 20 weeks, at 32 week
  Schedules for Clinical Assessment in Neuropsychiatry (SCAN), a semi-structured clinical interview with high reliability, is used to assess Axis I disorders. Diagnoses are assigned a clinical severity rating with a score of 0 (no symptoms attaining clinically significant severity) to 4 (severe interfering or disturbing in daily activity) as the clinical threshold for diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Shen-Ing Liu, Ph.D, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu SI, Chang CH, Lin CJ, Chen SC, Huang HC, Lin Y, Chang YH, Yeh HM, Lin IC, Wu SI. Modified dialectical behavior therapy-informed transdiagnostic intervention for emotional disorders: protocol for a randomized controlled trial. BMC Psychiatry. 2024 Nov 6;24(1):771. doi: 10.1186/s12888-024-06069-4. PMID 39506661